CLINICAL TRIAL: NCT06958120
Title: Analgesic Efficacy of Bilateral Ultrasound Guided Superficial Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block in Pediatric Patients Undergoing Corrective Cardiac Surgeries - A Randomized Controlled Study
Brief Title: Bilateral Ultrasound Guided Superficial Parasternal Intercostal Plane Block Versus Erector Spinae Plane Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Mahrous, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BLocks in pediatric cardiac op
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: CHD - Congenital Heart Disease
Keywords: CHD; Regional anaesthesia; Pain management
MeSH Terms: conditions — Heart Defects, Congenital; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial parasternal intercostal Plane block group (Experimental): This group will receive fentanyl infusion at a dose of (0.5μg/kg/h) all through the whole operation plus ultrasound guided bilateral superficial parasternal intercostal Plane block
  Interventions: Procedure: superficial parasternal intercostal Plane block
- Erecto-Spinea plane block group (Experimental): This group will receive fentanyl infusion at a dose of (0.5μg/kg/h) all through the whole operation plus Ultrasound guided bilateral Erecto-Spinea plane block
  Interventions: Procedure: Erecto spinea plane block

INTERVENTIONS:
Procedure: superficial parasternal intercostal Plane block — A high-frequency linear transducer was used to guide the insertion of a needle 2 cm lateral to the sternum. After identifying key anatomical structures, the needle was advanced in-plane into the pectointercostal fascial plane between the pectoralis major and internal intercostal muscle. Correct placement was confirmed with a saline injection, and then a local anesthetic (0.4 ml/kg of a 1:1 mix of bupivacaine 0.25% and lidocaine 1%) was injected bilaterally at the second and fourth ribs.
  Arms: Superficial parasternal intercostal Plane block group
Procedure: Erecto spinea plane block — Using ultrasound, a needle is inserted near the T5 vertebra into the plane beneath the erector spinae muscle. After confirming correct positioning with saline, a local anesthetic mixture is injected in the fascial plane.
  Arms: Erecto-Spinea plane block group

SUMMARY:
Group (A): This group will receive fentanyl infusion at a dose of (0.5μg/kg/h) all through the whole operation plus ultrasound guided bilateral superficial parasternal intercostal Plane block which will be done by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side3.

Group (B): This group will receive fentanyl infusion at a dose of (0.5μg/kg/h) all through the whole operation plus Ultrasound guided bilateral ESPB which will be done by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%) at each side .

DETAILED DESCRIPTION:
Preoperative assessment Premedication Monitoring General Anesthesia induction Arterial and Venous cannulation Fentanyl Infusion Giving block according to the group Intra operative recording of hemodynamics Post operative pain assessment

ELIGIBILITY:
Inclusion Criteria:

* RACHS-1: Categories 1, 2 and 3
* Patients undergoing corrective cardiac surgeries with midline sternotomy incision.
* Redo surgeries.

Exclusion Criteria:

* Patients whose parents or legal guardians refuse to participate.
* Preoperative mechanical ventilation.
* Preoperative inotropic drug infusion.
* Coagulopathy.
* Allergy to any of the studied drugs.
* Severe pulmonary hypertension (> 70 mmHg).

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | Immediately after admission to ICU then at 60 min, 2 hours, 4 hours, 8 hours and 12 hours postoperatively
  Pain was assessed by the pediatric observational 10-point scale "Face, Leg, Activity, Cry, Consolability (FLACC) pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Abu Al reesh hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2026
Access Criteria: Any